CLINICAL TRIAL: NCT05069948
Title: Delivery of Digital Cognitive Behavioural Therapy Following Concussion: HeadOn Feasibility Study
Brief Title: Delivery of Digital Cognitive Behavioural Therapy Following Concussion
Acronym: HEADON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/0151
Record Dates: First submitted 2021-09-27; First posted 2021-10-06 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2023-12

CONDITIONS: Concussion, Mild
Keywords: Cognitive behavioural therapy; Digital health; Traumatic brain injury
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HeadOn intervention (Experimental): Participants are given access to HeadOn - a web application that delivers a CBT programme to patients following concussion.
  Interventions: Other: HeadOn

INTERVENTIONS:
Other: HeadOn — HeadOn is a web application which takes the participant through a 5-stage CBT programme including: (i) understanding post-concussion symptoms; (ii) sleep after a concussion; (iii) lifestyle habits and exercise; (iv) managing negative thought patterns and (v) returning to baseline. The programme is delivered through a combination of weekly tasks (such as completing symptom diary, setting exercise goals and setting up a sleep time routine), audio/video media and reading material.

SUMMARY:
Concussion is common and patients can go on to suffer with a constellation of symptoms which impacts their functional outcome and quality of life. Patient provision with information about their concussion and subsequent follow-up is highly variable. The investigators have developed HeadOn - a web application that delivers a CBT programme to patients following concussion. In this study, the investigators would like to examine the feasibility of digitally delivering a course of CBT to patients following concussion.

DETAILED DESCRIPTION:
The HeadOn study is a prospective feasibility study of patients presenting to the Emergency Department (ED). Potentially eligible patients will be contacted by a member of the research team and their consent will be sought for participation. Those not recruited at presentation to the ED will be contacted by telephone, text or email within two weeks of their concussion date to seek their participation in the study, again by a member of the research team. After consenting, the participant will be taken through the registration process for the HeadOn program. For patients who are contacted after discharge they will be taken through registration process over the telephone or if preferable will be able to return to the ED to go over the process.

At registration the participant will be invited to complete a series of patient reported measures including the Rivermead post-concussion questionnaire, Pittsburgh Sleep Quality Index, PHQ9 questionnaire and FAST alcohol questionnaire within the HeadOn program. Alongside this, a series of researcher-led anonymised data points will be collected in a separate specially designed database including demographics, date of concussion, neurological and imaging findings which will all be collected from the medical notes and imaging reports. The HeadOn program runs for five weeks following which the participant will be invited to complete the same set of outcome measures. Alongside this, all the participant will be contacted (via telephone, text or email) by a member of the research team at week 5 to complete a further five measurements: Glasgow Outcome Score Extended, mHealth App Usability questionnaire, time to return to work and a healthcare utility questionnaire. Interested participants will be invited back within two months of enrolling in the study for a more detailed qualitative interviews about HeadOn. The study will recruit for a period of 6-months or up to 100 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years and older (no upper age limit)
* Presenting to the ED with a concussion
* Concussion defined as a traumatically induced alteration of mental status (either defined as loss of consciousness and/or amnesia)
* Patient is Glasgow Coma Scale score of 13-15 on initial presentation to the ED
* Patient needs to be able to start using HeadOn within 14 days of their head injury

Exclusion Criteria:

* Patients aged under 16 years old
* Patients requiring surgical management of their cranial injury
* Significant other associated injuries requiring hospitalisation (spinal injury, fractures, abdominal, cardiothoracic or vascular injuries)
* Does not have capacity to give consent
* Non-English speakers
* Patient in police custody or in prison

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimun Jamjoom, FRCS, Principal Investigator — University of Edinburgh
Locations (1):
- Edinburgh Royal Infirmary, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Annonymised study data will be made available on Edinburgh University's DataShare service
Time Frame: Data will be available for 5 years after completion of the study

REFERENCES:
- [Derived] d'Offay C, Ng XY, Alexander L, Grant A, Grahamslaw J, Pagliari C, Reed MJ, Carson A, Gillespie DC, Jamjoom AAB. A Digital Health Intervention for Concussion: Development and Clinical Feasibility Study. JMIR Form Res. 2023 Feb 1;7:e43557. doi: 10.2196/43557. PMID 36724010

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HeadOn Intervention
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HeadOn Intervention
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50

OUTCOME MEASURES:

1. Primary Outcome: Participant Compliance With HeadOn Program
Description: Degree of engagement of study participants with the HeadOn program. This was defined as whether the participant entered data into the HeadOn functionality (including symptom diary, sleep time setting, alcohol tracker, exercise day setting, thought diary and goal setter)
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Groups:
- HeadOn Cohort: Cohort of 50 study participants using HeadOn
Arm/Group | HeadOn Cohort
Number analyzed (Participants) | 50
Participants
  Symptom diary compliance | 45
  Non-compliance | 5

2. Secondary Outcome: mHealth App Usability Questionnaire
Description: The mobile Health App Usability Questionnaire (MAUQ) is a validated questionnaire that examine participants' attitudes to an mHealth intervention. MAUQ quantifies respondents' perceptions of the usability of a mobile health app using a range from 1 to 7. A score of 7 indicates a high degree of usability.
Time Frame: 5 weeks
Population: Only 29 (out of 50) participants responded to this questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HeadOn Cohort
Number analyzed (Participants) | 29
units on a scale | 6.1 (1.3)

3. Secondary Outcome: Rivermead Post-concussion Questionnaire
Description: The Rivermead Post-Concussion Symptom Questionnaire (RPQ) is a self-report scale to measure the severity of post-concussive symptoms following a Traumatic Brain Injury. It examines 16 post-concussion symptoms which are rates from 0 (no symptom) to 4 (severe symptom). This gives a range from 0 (o post-concussion symptoms) to 64 (severe post-concessional symptoms).
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeadOn Cohort
Number analyzed (Participants) | 22
score on a scale | 16 (13)

4. Secondary Outcome: PHQ9 Questionnaire
Description: The Patient Health Questionnaire (PHQ)-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Range include 0 (no depression) to 27 (severe depression).
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeadOn Cohort
Number analyzed (Participants) | 22
score on a scale | 8 (7)

5. Secondary Outcome: Glasgow Outcome Score Extended
Description: The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status. There are 8 categories that are denoted numerically as follows: Dead (1), Vegetative State (2), Lower Severe Disability (3), Upper Severe Disability (4), Lower Moderate Disability (5), Upper Moderate Disability (6), Lower Good Recovery (7), and Upper Good Recovery (8).
Time Frame: 5 weeks
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | HeadOn Cohort
Number analyzed (Participants) | 29
Score on a scale | 8 [4 to 8]

6. Secondary Outcome: Return to Work Rate
Description: Patient self reported outcome measure. Participants were contacted by telephone at the completion of HeadOn (5 weeks from registration) and asked the following question 'Have you returned to work?'. The outcome was dichotomous and was either coded as 'yes' or 'no' based on participant response. The measure was then reported as a return to work rate which was the percentage of participants who reported they had returned to work at the completion of HeadOn.
Time Frame: 5 weeks
Population: 25 participants responded to this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | HeadOn Cohort
Number analyzed (Participants) | 25
Participants | 10

7. Secondary Outcome: Healthcare Resource Utilisation
Description: Patient Self reported outcome measure. At completion of the HeadOn program (5 weeks from registration), the participants were contacted by telephone and were asked 'Have you sought healthcare professional support due to your post-concussion symptoms since you started using HeadOn?'. The outcome was a dichotomous outcome and was either coded as 'yes' or 'no'. The definition of healthcare professional included: returning to the emergency department, seeing family doctor, a neuropsychologist, physiotherapist or sports medicine doctor). The outcome measure was reported as the percentage of respondents who sought healthcare professional input while using HeadOn.
Time Frame: 5 weeks
Population: 29 participants responded to this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | HeadOn Cohort
Number analyzed (Participants) | 29
Participants | 10

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | HeadOn Intervention
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT05069948/Prot_SAP_000.pdf